CLINICAL TRIAL: NCT06966102
Title: Evaluating the Effect of Lidocaine Infusion Versus Magnesium Sulfate Infusion on Decreasing Total Fentanyl Requirements in Patients Undergoing Functional Endoscopic Sinus Surgeries: a Randomized Controlled Study
Brief Title: Lidocaine Infusion Versus Magnesium Infusion in Decreasing Fentanyl Requirements in Endoscopic Sinus Surgeries
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kareem Mohammed Assem Nawwar, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MS-15-2025
Record Dates: First submitted 2025-05-03; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Enhanced Recovery; Functional Endoscopic Sinus Surgery; Lidocaine; Magnesium Sulphate; Perioperative Pain
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group L (Active Comparator): Patients received 2 mg/kg/h lidocaine hydrocloride starting at induction of anesthesia and continuing until the end of surgery
  Interventions: Drug: Lidocaine group
- Group M (Active Comparator): Patients received magnesium sulphate 20 mg/kg/h starting at induction of anesthesia and continuing until the end of surgery
  Interventions: Drug: Magnesium group
- Group C (Sham Comparator): Patients received saline infusion starting at induction of anesthesia and continuing until the end of surgery
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Lidocaine group — 25ml of lidocaine hydrochloride 2% will be added to 25 ml of standard saline 0.9% solution in a 50ml syringe to be infused via a syringe pump. The resultant concentration will be 10mg/ml. According to the calculated study drug dose, each patient will receive 0.2ml/kg/h
  Arms: Group L
Drug: Magnesium group — a 50ml syringe will be filled with magnesium sulfate solution (100mg/ml) to be infused via a syringe pump. According to the calculated study drug dose, each patient will receive 0.2ml/kg/h
  Arms: Group M
Drug: Control group — a 50ml syringe will be filled with a standard saline 0.9% solution to be infused via a syringe pump. Each patient will receive 0.2ml/kg/h
  Arms: Group C

SUMMARY:
Enhanced recovery after ear, nose and throat surgery is based on multimodal and multidisciplinary perioperative interventions to decrease postoperative pain. Functional endoscopic sinus surgery is a surgical management for chronic rhinosinusitis. Although a common procedure, there is a lack of knowledge about perioperative pain and specific pain management after such a procedure. Most of recommendations given in guidelines for postoperative pain management in nasal surgery and sinus surgery are subsumed under head and neck surgery. Head and neck surgery is a wide field covering widely variable surgical procedures. So, postoperative pain management guidelines may not meet the requirements for pain management during and after endoscopic sinus surgery.

Various medications have been used to improve the surgical field and postoperative pain including intravenous clonidine, dexmedetomidine, lidocaine, and magnesium.

Lidocaine has been used considering its analgesic, immuno-modulating, and anti-inflammatory properties. The opioid sparing effect of lidocaine is supported by a high level of evidence. The effectiveness of lidocaine infusion in obtaining reduction of postoperative pain, gastrointestinal recovery time, postoperative nausea and vomiting, and shortening the hospital length of stay, was demonstrated principally in major gastro-intestinal surgery.

Magnesium sulfate is a good option in multimodal analgesia, as it stabilizes the cell membrane and intracytoplasmic organelles by mediating the activation of Na+-K+ ATPase and Ca++ ATPase enzymes, which have an important role in transmembrane ion exchange during the depolarization and repolarization phases. Moreover, magnesium inhibits the release of norepinephrine by blocking the N-type Ca++ channels at nerve endings.

Many studies were designed to prove the role of the analgesic effect of lidocaine and magnesium infusion. However, this is the first randomized controlled study to assess the effect of lidocaine infusion versus magnesium sulphate infusion on decreasing total fentanyl requirements in patients undergoing functional endoscopic sinus surgery.

This randomized controlled trial was designed to compare the efficacy of lidocaine hydrochloride infusion versus magnesium sulphate infusion in controlling perioperative pain in patients undergoing functional endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 60 years.
* Both genders.
* American society of Anesthesiologist (ASA) physical status I-II
* Scheduled for functional endoscopic sinus surgery under general anesthesia.

Exclusion Criteria:

* Patients with prolonged QT interval.
* Patients with renal disease.
* Patients with a history of allergy to lidocaine or magnesium sulfate.
* American Society of Anesthesiologists class higher than II.
* Patient refusal

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
intraoperative fentanyl consumption | for 5 hours starting from induction of general anesthesia
  total fentanyl consumption during surgery

SECONDARY OUTCOMES:
intraoperative mean arterial blood pressure | for 5 hours starting from induction of general anesthesia
  mean arterial blood pressure during surgery
Intraoperative heart rate | for 5 hours starting from induction of general anesthesia
  heart rate during surgery
Clarity of the surgical field | for 5 hours starting from induction of general anesthesia
  Clarity of the surgical field according to Fromme and Boezaart scale (grade 0 means no bleeding and grade 5 means High bleeding, so constant blood evacuation is needed)
Surgeon satisfaction | for 5 hours starting from induction of general anesthesia
  Surgeon satisfaction assessed at the end of the operation on a 5-point Likert satisfaction scale (grade 1 means Extremely dissatisfied and grade 5 means Extremely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Jehan Elkholy, M.D., Study Chair — Cairo University; Kareem MA Nawwar, M.D., Study Director — Cairo University; Dina M Mohamed, M.D., Study Director — Cairo University; Dalia G Abdel Nasser, M.B.B.Ch., Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt